CLINICAL TRIAL: NCT04070391
Title: Vitamin B6 Supplementation and Mood States in College Women Taking Oral Contraceptives
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Principal Investigator, Carol Johnston, Professor and Associated Dean, Arizona State University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: VitB6OC
Record Dates: First submitted 2019-07-01; First posted 2019-08-28 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Depression
Keywords: vitamin B6; contraception; depression
MeSH Terms: conditions — Depression | interventions — Vitamin B 6

STUDY DESIGN:
Intervention Model Description: At the start of the trial, participants are instructed to take the provided pills once daily for four weeks. For weeks 5-8, participants will not take any pills (the washout period). Daily pill consumption will resume during weeks 9-12 (the crossover treatment). Participants are their own control in this crossover trial.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The student investigator (only investigator interacting with participants) and all participants were blinded to the active supplement.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vitamin B6 (Experimental): One pill (100 mg) ingested daily for 4 weeks.
  Interventions: Dietary Supplement: vitamin B6
- control (Placebo Comparator): One vinegar pill ingested daily for 4 weeks
  Interventions: Other: control

INTERVENTIONS:
Dietary Supplement: vitamin B6 — oral administration
  Arms: vitamin B6
Other: control — oral administration
  Arms: control

SUMMARY:
Purpose of Study The purpose of this crossover study was to determine how vitamin B6 supplementation impacts mood states in college age (18-25 y) women that use oral contraceptives, in comparison to a placebo treatment.

Hypothesis Daily supplementation of vitamin B6 (100 mg) over a 4-week period will improve mood states in college age women (18-25 y) with marginal vitamin B6 status that use oral contraceptives, compared to the placebo treatment.

DETAILED DESCRIPTION:
This study is a 12-week, randomized, double-blinded crossover trial. After eligibility is confirmed through prescreening and onsite screening assessments (screening visit; ~30 minutes), participants will sign the consent form and enter the trial. Participants are stratified by age, BMI, and length of oral contraceptive use and randomized by a coin flip into the experimental group (B6 supplement) or control group (low does vinegar pill). Participants will visit the test site in the fasted state (no food or drink with the exception of water for 10 hours) on 4 occasions (pre and post weeks 1-4 and pre and post weeks 9-12) These visits are approximately 30 minutes long. At the start of the trial, participants are instructed to take the provided pills once daily for four weeks. For weeks 5-8, participants will not take any pills (the washout period). Daily pill consumption will resume during weeks 9-12 (the crossover treatment). Participants are their own control in this crossover trial.

All participants are instructed to maintain their normal exercise and eating patterns consistently throughout the duration of the 12-week study. Additionally, participants are instructed not to start any new medications or nutritional/herbal supplements. To promote compliance, participants will have a calendar to check off each day that the pills are consumed during the study.

Anthropometric data are collected and fasting blood draws are performed at weeks 0, 4, 9 and 12. Fasting blood samples will be tested for B6 and associated metabolites. Additionally, mood assessments, including the Profile of Mood States and the Beck Depression Inventory will be administered at weeks 0, 4, 9 and 12.

ELIGIBILITY:
Inclusion Criteria:

* Female who has taken a combined oral contraceptive (estrogen with progestin) consistently for at least one year
* Healthy by self-report; no active disease state, depressive state, or prescription medication use (exception: OC)
* 18-25 years of age
* Nonsmoking
* Not pregnant or lactating if female
* Not a regular user of supplements aside from multivitamin/mineral supplement
* Dietary B6 at or below the RDA (1.3 mg/day)
* Not vegetarian/vegan
* Not a competitive athlete

Exclusion Criteria:

* Unwilling to take a vitamin supplement or placebo daily as prescribed during the 12 week study
* Unable to meet with investigators and provide a fasting blood sample on 4 occasions over a 12 week period

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — use of oral contraception
Enrollment: 8 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Depression | change from baseline to week 4
  Beck Depression Inventory: a twenty-one question measure (item score, 0-3); the highest possible total for the whole test is sixty-three.

SECONDARY OUTCOMES:
Plasma vitamin B6 | change from baseline to week 4
  ELISA assay

CONTACTS AND LOCATIONS:
Overall Officials: Susan Metosky, MS, Study Director — Institutional Review Board
Locations (1):
- Arizona State University, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No